CLINICAL TRIAL: NCT03231982
Title: A Randomized, Double-blind, Multi-center, Phase Ⅳ Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety Between Amlodipine Besylate/Candesartan Cilexetil Combination Tablets and Co-administration of Amlodipine Besylate and Candesartan Cilexetil in Patients With Essential Hypertension
Brief Title: Study to Confirm the Efficacy and Safety of Fixed-dose Combinations of Amlodipine and Candesartan
Acronym: MACH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_CCA_401
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Fixed-Dose combination of Candesartan cilexetil 8mg and Amlodipine 5mg(or Fixed-Dose combination of Candesartan cilexetil 16mg and Amlodipine 5mg), once a day for 8 weeks
  Interventions: Drug: Group I
- Group II (Active Comparator): Candesartan cilexetil 8mg and Amlodipine 5mg(or Candesartan cilexetil 16mg and Amlodipine 5mg), once a day for 8 weeks
  Interventions: Drug: Group II

INTERVENTIONS:
Drug: Group I — Machkhan Tab. 8/5 mg + Atacan Tab. 8 mg placebo + Norvasc Tab. 5 mg placebo for 8 weeks or Machkhan Tab. 16/5 mg + Atacan Tab. 16 mg placebo + Norvasc Tab. 5 mg placebo for 8 weeks
  Other Names: Machkhan Tab. 8/5 mg(or Machkhan Tab. 16/5 mg)
  Arms: Group I
Drug: Group II — Atacan Tab. 8 mg + Norvasc Tab. 5 mg + Machkhan Tab.8/5 mg placebo for 8 weeks or Atacan Tab. 16 mg + Norvasc Tab. 5 mg + Machkhan Tab.16/5 mg placebo for 8 weeks
  Other Names: Atacan Tab. 8 mg(or Atacan Tab. 16 mg), Norvasc Tab. 5 mg
  Arms: Group II

SUMMARY:
To evaluate the efficacy and safety of amlodipine besylate and candesartan cilexetil administered in a fixed-dose combination tablet versus co-administered as their separate formulations in patients with essential hypertension who have shown inadequate response on monotherapy of amlodipine or candesartan cilexetil or who are with blood pressure adequately controlled by co-administration of amlodipine besylate and candesartan cilexetil single agents

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female aged 19 to 75 years
2. Diagnosed with essential hypertension

   Patients with essential hypertension meeting one of the following two inclusion criteria:

   2.1. Patients with essential hypertension who have shown inadequate response (mean siSBP ≥ 140 mmHg or mean siDBP ≥ 90 mmHg) to treatment with amlodipine or candesartan cilexetil.

   2.2. Patients with essential hypertension with blood pressure adequately controlled by co-administration of amlodipine besylate and candesartan cilexetil (mean siSBP < 140 mmHg and mean siDBP < 90 mmHg).
3. Voluntarily consented to participate in the study and signed the informed consent form after receiving the explanation of the objectives, methods and effects of the study.

Exclusion Criteria:

1. The difference in blood pressure between the selected arm versus non-selected arm is ≥ 20 mmHg for siSBP and ≥ 10 mmHg for siDBP at Visit 1 (screening).
2. Blood pressure taken at screening and randomization is ≥ 180 mmHg for siSBP or ≥ 110 mmHg for siDBP.
3. Diagnosed with secondary hypertension or suspected of secondary hypertension [e.g., renovascular disease, adrenal medullary and cortical hyperfunction, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc.]
4. Patients with symptomatic orthostatic hypertension (the difference in the blood pressures between measured at supine position and measured at standing position is ≥ 20 mmHg for siSBP and ≥ 10 mmHg for siDBP)
5. Diagnosis of type 1 diabetes mellitus (DM) or uncontrolled DM (patients on insulin therapy or with HbA1c > 9%)
6. Patients with severe cardiac conditions: heart failure (NYHA Class 3 or 4), history of ischemic cardiac disease (unstable angina, myocardial infarction), peripheral vascular diseases, percutaneous transluminal angioplasty or coronary artery bypass graft within recent 6 months.
7. Patients with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically significant arrhythmia at the discretion of the investigator
8. Patients with hypertrophic occlusive myocardiopathy, severe occlusive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve stenosis
9. History of cardiogenic shock
10. Presence of severe cerebrovascular disorders (diagnosis of stroke, cerebral infarction or cerebral hemorrhage within recent 6 months)
11. History or current evidence of wasting, autoimmune (such as rheumatoid arthritis and systemic lupus erythematosus) or connective tissue diseases
12. Known diagnosis of moderate or malignant retinopathy (including retinal hemorrhage, visual disturbance and retinal microaneurysm within 6 months)
13. Patients with surgical or medical intestinal diseases or having received surgeries that could interfere with drug absorption distribution, metabolism and elimination
14. History of malignancy including leukemia and lymphoma within recent 5 years except for localized basal cell carcinoma of the skin)
15. Patients with any inflammatory diseases requiring chronic anti-inflammatory therapy
16. Renal failure on dialysis
17. Laboratory abnormalities as follows:

    * AST or ALT >2 x upper limit of normal (ULN)
    * Serum creatinine > 1.5 x ULN
    * Serum potassium < 3.5 mmol/L or >5.5 mmol/L
18. Needs for co-administration of non-study antihypertensive agents or contraindicated medications during the study
19. History of hypersensitivity to ARBs or dihydropyridines
20. History of angioedema to treatment with ACE inhibitors or ARBs
21. Pregnant or lactating women and female volunteers of childbearing potential (except for women who are surgically sterile) who are not willing to use an adequate method of contraception (oral contraceptives, intrauterine device, condom, etc.) during the study. Women of childbearing potential who are not surgically sterile will be allowed to participate in the study only if they have negative pregnancy test at Visit 1 (screening) and should continue to use medically acceptable method of contraception (basic body temperature method and rhythm method will not be allowed). Women with no menses for ≥ 12 months will be considered as postmenopausal state and method of contraception using hormonal contraception such as oral contraceptive should be initiated from or prior to the screening.
22. History of drug or alcohol abuse within recent 1 year
23. Patients having received any other investigational product within recent 12 weeks
24. Conditions which render a subject ineligible for the study at the discretion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in sitting Systolic Blood Pressure(siSBP) from baseline after 8 weeks of treatment | Week 8
  For change in siSBP from baseline after 8 weeks of treatment, the mean, standard deviation, median, minimum and maximum will be presented by treatment arm.
  The LS mean change in siSBP from baseline after 8 weeks of treatment adjusted for baseline siSBP and its standard error will be presented by treatment arm. Non-inferiority test will be conducted using ANCOVA including change in siSBP from baseline after 8 weeks of treatment as response variable and baseline siSBP and treatment arm as independent variables. Amlodipine besylate/candesartan cilexetil combination tablet will be considered non-inferior to co-administration of amlodipine besylate and candesartan cilexetil if the lower bound of 2-sided 95% CI for the LS mean of difference in siSBP change between the treatment arms is greater than -5.

SECONDARY OUTCOMES:
Change in siSBP from baseline after 4 weeks of treatment | Week 4
  For change in siSBP from baseline after 4 weeks of treatment, the mean, standard deviation, median, minimum and maximum will be presented by treatment arm.
  The LS mean change in siSBP from baseline after 4 weeks of treatment adjusted for baseline siSBP and its standard error will be presented by treatment arm. Non-inferiority test will be conducted using ANCOVA including change in siSBP from baseline after 4 weeks of treatment as response variable and baseline siSBP and treatment arm as independent variables. Amlodipine besylate/candesartan cilexetil combination tablet will be considered non-inferior to co-administration of amlodipine besylate and candesartan cilexetil if the lower bound of 2-sided 95% CI for the LS mean of difference in siSBP change between the treatment arms is greater than -5.
Change in siDBP from baseline after 4 and 8 weeks of treatment | Week 4 and Week 8
  For change in siDBP from baseline after 4 and 8 weeks of treatment, the mean, standard deviation, median, minimum and maximum will be presented by treatment arm.
  The LS mean change in siSBP from baseline after 4 and 8 weeks of treatment adjusted for baseline siDBP and its standard error will be presented by treatment arm. Non-inferiority test will be conducted using ANCOVA including change in siDBP from baseline after 4 and 8 weeks of treatment as response variable and baseline siDBP and treatment arm as independent variables. Amlodipine besylate/candesartan cilexetil combination tablet will be considered non-inferior to co-administration of amlodipine besylate and candesartan cilexetil if the lower bound of 2-sided 95% CI for the LS mean of difference in siSBP change between the treatment arms is greater than -5.
Proportion of subjects with siDBP < 90 mmHg and siSBP <140 mmHg after 8 weeks of treatment | Week8
  The frequency and percentage of subjects with siDBP < 90 mmHg and the frequency and percentage of subjects with siSBP < 140 mmHg after 8 weeks of treatment will be presented by treatment arm. Additionally, the frequency and percentage of subjects with both siDBP < 90 mmHg and siSBP <140 mmHg after 8 weeks of treatment will be presented by treatment arm. The difference in proportion between treatment arms will be tested using the χ2 test or Fisher's exact test.

OTHER OUTCOMES:
Adverse events | Baseline, Week 4 and Week 8
  All patients treated with the investigational product will be included in the safety analyses. For adverse events, adverse drug reactions and serious adverse events, the number of subjects experiencing the events or reactions, 95% 2-sided CI, incidence rate, and number of the events or reactions will be presented by treatment arm. The difference in the incidence between the treatment arms will be tested using the χ2 test or Fisher's exact test. The incidence and percentage of events by severity, causality, actions taken and outcome will be presented by treatment arm.
  All AEs will be coded per system organ class (SOC) and preferred term (PT) using the MedDRA; for each coded event, the number and percentage of subjects and the number of cases will be summarized by treatment arm. In addition, for each coded event, the number and percentage of subjects by severity, causality, actions taken and outcome will be presented by treatment arm.
Clinical laboratory tests | Baseline, Wee4 and Week 8
  For continuous variables in clinical laboratory test items, the mean, standard deviation, minimum and maximum of baseline value, post-baseline values and change form baseline to post-baseline will be presented by treatment arm. The difference in change from baseline to post-baseline between treatment arms will be tested using the unpaired t-test or Wilcoxon's rank sum test depending on the normality. The intra-arm change from baseline to post-baseline will be tested using the paired t-test or Wilcoxon's signed rank test depending on the normality. For categorical variables, the shift table for frequency and percentage will be presented. The difference in the percentage of subjects whose test results changed from 'normal' to 'abnormal' between treatment arms will be tested using the χ2 test or Fisher's exact test. The intra-arm change from baseline to post-baseline will be tested using the McNemar's test.
Electrocardiogram (ECG) | Screening and Week 8
  For each ECG parameters at baseline and post-baseline, the shift table will be presented with frequency and percentage. The difference in the percentage of subjects whose ECG results changed from 'clinically insignificant' to 'clinically significant' between treatment arms will be tested using the χ2 test or Fisher's exact test. The intra-arm change from baseline to post-baseline will be tested using the McNemar's test.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Cardiovascular Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No